CLINICAL TRIAL: NCT06949358
Title: A Long-Term Follow-up Study to Evaluate Safety and Tolerability of Olipudase Alfa in Patients Who Completed the DFI12712 or the LTS13632 Study in France
Brief Title: A Study to Evaluate Safety and Tolerability of Olipudase Alfa in Pediatric and Adult Participants With Acid Sphingomyelinase Deficiency (ASMD) Who Completed the DFI12712 or the LTS13632 Study in France
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTA17397; 2024-515304-39 (Registry Identifier: CTIS); 2021-004109-39 (EudraCT Number)
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Niemann-Pick Disease
MeSH Terms: conditions — Niemann-Pick Diseases | interventions — olipudase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- GZ402665 (Experimental): Olipudase alfa administered intravenously every 2 weeks
  Interventions: Drug: Olipudase alfa

INTERVENTIONS:
Drug: Olipudase alfa — Pharmaceutical form:Powder for concentrate for solution for infusion-Route of administration:intravenous infusion
  Other Names: GZ402665

SUMMARY:
This is an open-label study to evaluate safety and tolerability and provide enzyme replacement therapy (ERT) with olipudase alfa to patients with acid sphingomyelinase deficiency (ASMD) who completed the DFI12712 or the LTS13632 Study in France until olipudase alfa reimbursement is granted in France.

Study and treatment duration:

The period between the patient's completion of Study DFI12712 or LTS13632 and olipudase alfa reimbursement is available in France.

In case reimbursement will not be obtained, this study will end 5 years after starting.

Visit frequency: every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The patient has completed Study DFI12712 (ASCEND) or LTS13632 in France
* The patient must provide signed, informed consent prior to performing any study-related procedures.
* The patient is willing to comply with the clinical protocol.
* The patient, if female and of childbearing potential, must have a negative pregnancy test result [urine beta-human chorionic gonadotropin (β-HCG)] at enrollment.
* Sexually active female patients of childbearing potential and male patients are required to practice true abstinence in line with their preferred and usual lifestyle or to use 2 acceptable effective methods of contraception for the entire duration of the treatment period and for at least 28 days after receiving the last study drug dose.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Any patient who has not participated in the Study DFI12712 or the Study LTS13632
* A patient who experienced any systemic hypersensitivity reactions to olipudase alfa in Study DFI12712 or Study LTS13632 which, in the opinion of the Investigator, could indicate that treatment continuation may present an unreasonable risk.
* The patient, in the opinion of the Investigator, is unable to adhere to the requirements of the study.
* The patient is unwilling or unable to abstain from alcohol for 1 day prior to and 3 days after each olipudase alfa infusion for the duration of the treatment period.
* Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalized.
* The patient is concurrently participating in another clinical study of investigational treatment.
* Any of the following medical conditions:
* The patient has any new condition or worsening of an existing condition which, in the opinion of the Investigator, would make the patient unsuitable for enrollment or could interfere with the patient's participating in or completing the study.
* Requirement for recurrent dose adjustment of anticoagulation treatment over the last 6 months.
* Pregnancy or breastfeeding.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) / serious adverse events (SAEs) | Baseline to approximately 5 years

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Investigational Site Number : 2500002, Bron
  - Investigational Site Number : 2500001, Paris

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org